CLINICAL TRIAL: NCT03367754
Title: A Randomized, Double-Blind, Placebo-Controlled Study of a Single Dose of Pembrolizumab in HIV-Infected Patients
Brief Title: A Single Dose of Pembrolizumab in HIV-Infected People
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with subject recruitment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180013; 18-CC-0013
Record Dates: First submitted 2017-12-08; First posted 2017-12-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Human Immunodeficiency Virus
Keywords: Immunotherapy; Immunologic Non-Responder; Immunologic Response; Randomized; PD-1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Pembrolizumab (Experimental): Participants with HIV and CD4+ of 100-350 cells/mm^3 received a single dose of Pembrolizumab 200 mg via intravenous (IV) infusion.
  Interventions: Drug: Pembrolizumab
- Placebo (Placebo Comparator): Participants with HIV and CD4+ of 100-350 cells/mm^3 received a single dose of Placebo via intravenous (IV) infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Single dose of Placebo given via intravenous (IV) infusion.
  Arms: Placebo
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (immunoglobulin [Ig] G4 kappa isotype) that binds to PD-1, thus blocking the receptor from binding with its ligands. Single dose of Pembrolizumab 200 mg given via intravenous (IV) infusion.
  Arms: Drug: Pembrolizumab

SUMMARY:
Background:

Human immunodeficiency virus (HIV) attacks the immune system. Some people with HIV have a low CD4+ T-cell count despite taking antiviral medicines that control HIV replication. These cells fight disease, so a low count makes it easier for people to become sick. Researchers want to see if a new drug can improve the immune system, including T cells. The drug is called pembrolizumab

Objective:

To see if pembrolizumab is safe to use in people with HIV who have a low CD4+ T cell count despite taking medicines that control HIV replication, and to see if it strengthens the immune system.

Eligibility:

People age 18 years or older with HIV who are taking antiretroviral drugs as treatment, have blood HIV levels below detection limits of commercial assays, and have a low CD4+ T-cell count (below 350 cells/mm3).

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Heart, blood, and urine tests

Sexually active participants must use 2 kinds of birth control.

Participants will have leukapheresis. Blood will be removed through a needle in one arm. A machine will remove white blood cells. The rest of the blood will be returned into the other arm.

Participants will have a baseline visit. They will have blood tests. They may have a pregnancy test.

A needle will insert a thin plastic tube (IV) into an arm vein. The participants will get the study drug or a placebo through the IV for 30 minutes. They will be watched for a couple hours after.

Participants will have 11 follow-up visits over the next 48 weeks. They will have a physical exam, vital signs, medical review, and blood tests.

Participants may have another leukapheresis.

Participants will be called every 12 weeks after their last follow-up visit to talk about how they feel and their health. Participation ends after the week 96 phone call.

DETAILED DESCRIPTION:
A subset of HIV-infected patients, those with poor immunologic response to combined antiretroviral therapy (CD4+ T-cell count of less than 300-350 cells/mm^3) despite control of viremia, are at increased risk for both HIV-related and non-HIV-related complications compared to immunologic responders. Thus, novel approaches for treating HIV infection are needed to facilitate management of this patient population.

One potential drug target for HIV treatment is the T-cell receptor PD-1. Binding of PD-1 to its ligands, PD-L1 and PD-L2, inhibits proliferation of T cells and production of cytokines. This naturally serves to dampen potentially harmful excessive immune responses. Upregulation of PD-1 and/or its ligands can be observed in tumors and people with chronic viral infection, including HIV. This upregulation can inhibit T-cell immune surveillance, which may result in tumor growth or poor control of infection.

Pembrolizumab is an IgG4 kappa monoclonal antibody that binds to PD-1, thus blocking the receptor from binding with its ligands. In cancer indications, inhibition of PD-1 induces an antitumor immune response, which in turn reduces tumor growth. The Food and Drug Administration has approved pembrolizumab for treatment of unresectable or metastatic melanoma, non-small cell lung cancer, head and neck squamous cell carcinoma, and other cancers. Similarly, in animal models of HIV and in vitro studies, PD-1 blockade was associated with a decrease in viral load and an increase in CD8+ T cells. A clinical trial to examine the effects of PD-1 inhibition by pembrolizumab on HIV infection is thus supported by the data.

The purpose of this study is to evaluate, in a randomized, double-blind, placebo-controlled study, the safety and tolerability of a single dose of pembrolizumab in HIV-infected participants who have controlled viremia with a low T-cell count (> 100 cells/mm3 and less than or equal to 350 cells/mm^3). Study participants will be followed for 96 weeks after receiving the study drug and will be assessed for adverse events, CD4+ and CD8+ T-cell counts, PD-1 expression, CD8+ T-cell anti-HIV activity, and viral load. If a single dose of pembrolizumab appears to be safe and tolerable, then larger multi-dose and efficacy studies can be planned.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Greater than or equal to 18 years of age.
* Documented HIV-1 infection (eg, positive standard enzyme-linked immunosorbent assay or rapid HIV-1/HIV-2 antibody test with a confirmatory test such as western blot, or documentation of repeated HIV RNA of > 1000 copies/mL). Outside documentation will be acceptable.
* Absolute neutrophil count > 1000/microliter.
* Platelet count > 125,000/microliter.
* Hemoglobin > 10 g/dL.
* Aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 1.1 times the upper limit of normal (ULN). Total bilirubin < 1.1 x ULN (unless participant is taking atazanavir or has Gilbert syndrome).
* Calculated creatinine clearance (estimated glomerular filtration rate) greater than or equal to 60 mL/min/1.73 m2.
* Thyroid-stimulating hormone (TSH) and adrenocorticotropic hormone (ACTH) within normal limits. If TSH is not within normal limits then the participant may be eligible if thyroxine (T4) is within normal limits. Participants will not be excluded if they are on a stable dose of replacement thyroid medication; dose may be adjusted as needed.
* No significant underlying pulmonary, cardiac, renal, or hepatic disease, as defined by a need for drug treatment or ongoing physician care.
* Under the care of a primary care physician.
* Willing to comply with study requirements and procedures including storage of biological specimens for future use in medical research.
* Willing to allow genetic testing.
* Able to provide informed consent.
* Participants of reproductive potential must agree to not become pregnant or to impregnate a partner beginning 30 days before the dose of pembrolizumab through 120 days post dose.

Participants must meet criteria for INR, defined as follows:

1. Has been on a cART regimen for at least 12 months and on a stable regimen for at least 4 weeks.
2. Has HIV suppression, defined as viral load < 40 copies/mL, and documented suppression (below detection limits of the utilized assay) for at least 12 months. A viral load of < 500 copies/mL once in the year preceding screening will be allowed if there is documentation of a viral load < 40 copies/mL on subsequent testing and at screening.
3. CD4+ T-cell count > 100 cells/mm3 and less than or equal to 350 cells/mm3.

EXCLUSION CRITERIA:

Females who are pregnant or breastfeeding.

Has used an investigational drug agent or investigational device within 12 weeks of baseline.

Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.

Known allergy to any component of the pembrolizumab formulation.

Systemic steroid therapy or other immunosuppressive therapy in the 3 months prior to enrollment (Inhaled or topical corticosteroids are permitted).

Has used an immunotherapeutic agent within 6 months of baseline.

Plans to receive any vaccine within 16 weeks of receiving pembrolizumab.

Has active autoimmune disease or a history of autoimmune disease that has required systemic treatment (eg, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, T4) is not considered a form of systemic treatment.

Has known history of, or any evidence of active, non-infectious pneumonitis.

Malignancy requiring systemic therapy, or a history of malignancy that required systemic therapy within the past 5 years. However, cutaneous basal cell carcinoma or cutaneous Kaposi sarcoma not requiring systemic therapy will not be exclusionary.

Has known active hepatitis B (HBV) or potential for HBV reactivation (eg, hepatitis B surface antigen [HBS] reactive, HBV DNA positive, or isolated anti-core antibody positive; individuals who are anti-HBS antibody positive with or without anti-core Ab are eligible).

Has known active hepatitis C (HCV; eg, HCV RNA [qualitative] is detected). Patients who have sustained virologic response (SVR) to anti-HCV treatment are eligible if at least 24 weeks have passed since achieving SVR.

Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

History or other clinical evidence of:

1. Significant or unstable cardiac disease
2. Significant pulmonary disease
3. Severe illness, chronic liver disease, malignancy, immunodeficiency other than HIV, active systemic infection (other than HIV) requiring therapy.

Opportunistic infection requiring maintenance therapy, including toxoplasmosis, fungal infections other than candida (eg, cryptococcosis, histoplasmosis, coccidioidomycosis), atypical mycobacterial infection. Secondary Pneumocystis, candida, and HSV prophylaxis will be permitted.

Active or history of tuberculosis (TB), or positive TB QuantiFERON Gold test.

Known osteoporosis or diabetes mellitus.

Hemoglobin A1c > 6%.

Fasting triglyceride > 300 mg/dL.

Any condition that, in the opinion of the investigator, would make the participant unsuitable for the study.

Co-enrollment in other trials is restricted, other than enrollment on observational studies or expanded access studies for antiretroviral agents, during the first 48 weeks of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study will be shared for future research as follows:
  Identified data in the Biomedical Translational Research Information System (BTRIS; automatic for activities in the CC).
  De-identified or identified data with approved outside collaborators under appropriate agreements.
  Through publication and/or public presentations.
  Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as a cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Time Frame: Data will be shared at the time of publication.
Access Criteria: Identified data in the Biomedical Translational Research Information System (BTRIS; automatic for activities in the CC).

REFERENCES:
- [Background] Gay CL, Bosch RJ, Ritz J, Hataye JM, Aga E, Tressler RL, Mason SW, Hwang CK, Grasela DM, Ray N, Cyktor JC, Coffin JM, Acosta EP, Koup RA, Mellors JW, Eron JJ; AIDS Clinical Trials 5326 Study Team. Clinical Trial of the Anti-PD-L1 Antibody BMS-936559 in HIV-1 Infected Participants on Suppressive Antiretroviral Therapy. J Infect Dis. 2017 Jun 1;215(11):1725-1733. doi: 10.1093/infdis/jix191. PMID 28431010
- [Background] Day CL, Kaufmann DE, Kiepiela P, Brown JA, Moodley ES, Reddy S, Mackey EW, Miller JD, Leslie AJ, DePierres C, Mncube Z, Duraiswamy J, Zhu B, Eichbaum Q, Altfeld M, Wherry EJ, Coovadia HM, Goulder PJ, Klenerman P, Ahmed R, Freeman GJ, Walker BD. PD-1 expression on HIV-specific T cells is associated with T-cell exhaustion and disease progression. Nature. 2006 Sep 21;443(7109):350-4. doi: 10.1038/nature05115. Epub 2006 Aug 20. PMID 16921384
- [Derived] Henderson LJ, Reoma LB, Kovacs JA, Nath A. Advances toward Curing HIV-1 Infection in Tissue Reservoirs. J Virol. 2020 Jan 17;94(3):e00375-19. doi: 10.1128/JVI.00375-19. Print 2020 Jan 17. PMID 31694954
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-CC-0013.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were enrolled on the study. Three participants were screen failure and one participants withdrew prior to start of study.
Period: Overall Study
Arm/Group | Drug: Pembrolizumab | Placebo
Started | 6 | 1
Completed | 6 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 6 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Either Grade 2 or Higher Autoimmune Events and Grade 3 or Higher Adverse Events
Description: Participants with either grade 2 or higher autoimmune events requiring corticosteroid therapy or grade 3 or higher adverse events that are possibly, probably, or definitely related to intervention. The severity of each adverse event was graded according to the "Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events".
  Grade 2: Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for ≤ 24 hrs.
  Grade 3: Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death
Time Frame: Up to 48 weeks from start of intervention
Population: Analysis included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants with HIV and CD4+ of 100-350 cells/mm^3 receive a single dose of Placebo via intravenous (IV) infusion.
Arm/Group | Drug: Pembrolizumab | Placebo
Number analyzed (Participants) | 6 | 1
Participants
  Grade 2 or higher autoimmune events requiring corticosteroid therapy | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 96 weeks from administration of intervention
Arm/Group | Drug: Pembrolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Pembrolizumab (N=6) | Placebo (N=1)
Chest pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: Pembrolizumab (N=6) | Placebo (N=1)
Coronary artery disease (Cardiac disorders) | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Vitreous floaters (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Cyst (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gonorrhoea (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 5 | 0
Blood corticotrophin abnormal (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 3 | 1
Blood phosphorus decreased (Investigations) | 2 | 0
Blood sodium increased (Investigations) | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 5 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Low density lipoprotein increased (Investigations) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated due to difficulty with participant recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03367754/Prot_SAP_000.pdf